CLINICAL TRIAL: NCT00769860
Title: Safety and Tolerability Trial of Arimoclomol for Sporadic Inclusion Body Myositis
Brief Title: Arimoclomol in Sporadic Inclusion Body Myositis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Richard Barohn, MD (Other)
Responsible Party: Sponsor-Investigator, Richard Barohn, MD, Gertrude and Dewey Zeigler Professor of Neurology and Chair, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10656
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-11

CONDITIONS: Inclusion Body Myositis
Keywords: myositis; IBM; inclusion body myositis
MeSH Terms: conditions — Myositis, Inclusion Body; Myositis | interventions — arimoclomol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Arimoclomol
  Interventions: Drug: Arimoclomol
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Arimoclomol — Arimoclomol 100 mg TID for 4 months
  Arms: 1
Other: Placebo — Placebo for 4 months
  Arms: 2

SUMMARY:
Inclusion body myositis (IBM) is the most common progressive and debilitating muscle disease beginning in persons over 50 years of age. This study will assess the safety and tolerability of Arimoclomol in IBM as compared to placebo over 4 months of treatment.

DETAILED DESCRIPTION:
IBM is a chronic disorder in which muscles become inflamed (swollen) and cause muscle weakening. The cause is unknown. There is new evidence to suggest that the pathology in IBM results from cellular changes induced by a variety of stressful events and diseases. In response to these stressful events the body's normal response is to increase the levels of Heat Shock Proteins (HSP) to help counteract and stop these cellular changes. In people with IBM this increase does not appear sufficient enough to reverse these toxic cellular changes. Arimoclomol causes the body to make more of this HSP protein. By increasing HSP levels in IBM patients we hope to reverse the toxic cellular changes that might be responsible for the pathology of IBM.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for definite or probable IBM (Griggs 1995)
* Muscle function adequate for quantitative muscle testing
* Age > 50 years
* Women must be postmenopausal or status post hysterectomy
* For any patient currently taking medication for IBM, they must remain on current dosage for the extent of the study and last dosage change must be > 30 days previous to enrollment

Exclusion Criteria:

* Presence of any one of the following medical conditions: diabetes mellitus or patients taking anti-diabetic medications, chronic infection, chronic renal insufficiency, cancer other than skin cancer less than 5 years previously, multiple sclerosis or prior episode or central nervous system demyelination, or other chronic serious medical illnesses
* Presence of any of the following on routine blood screening: WBC < 3000, platelets < 100,000, hematocrit < 30%, BUN > 30 mg%, creatine > 1.5 mg%, symptomatic liver disease with serum albumin < 3 g/dl, PT or PTT > upper range of control values
* Women who are pregnant or lactating
* History of non-compliance with other therapies
* Coexistence of other neuromuscular disease
* Drug or alcohol abuse within the last 3 months
* Inability to give informed consent
* Known bleeding disorder
* Use of potentially renal toxic drugs
* Prior difficulties with local anesthetic

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- University of Kansas Medical Center, Kansas City, Kansas, United States
- University College London, MRC Centre for Neuromuscular Disease, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matched placebo pills, 100 mg TID for 4 months
Period: Overall Study
Arm/Group | Arimoclomol | Placebo
Started | 16 | 8
Month 4 | 16 | 8
Month 8 | 14 | 8
Completed | 14 | 8
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arimoclomol | Placebo | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.85 (7.86) | 68.83 (6.70) | 66.84 (7.49)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 12 | 5 | 17
Region of Enrollment [Number; unit: participants]
  United States | 8 | 4 | 12
  United Kingdom | 8 | 4 | 12
Inclusion Body Myositis-Functional Rating Scale (IBMFRS) Score [Mean (Standard Deviation); unit: units on a scale] — The questionnaire has 10 questions. The maximum score is 40. The higher the score the better the functional status of the patient.
  units on a scale | 27.5 (7.0) | 24.6 (5.1) | 26.6 (6.4)
Manual Muscle Testing (MMT) Score [Mean (Standard Deviation); unit: units on a scale] — The MMT score range is 0-5. A score of 0 is the lowest and represents no visible or palpable contraction. A score of 5 is the highest and represents full range of motion against gravity, maximul resistance.
  units on a scale | 4.2 (0.5) | 3.6 (1.5) | 4.2 (0.4)
Maximum Isometric Voluntary Contraction Testing (MVICT) Score [Mean (Standard Deviation); unit: newtons] — Measured MVICT using the Quantitative Muscle Assessment (QMA) system designed by Computer Source, Atlanta, GA. The system uses an adjustable cuff to attach the patient's arm or leg to an inelastic strap that is connected to force transducer with a load of 0.5 to 1,000 Newtons. Maximum force is recorded.
  newtons | 130.4 (70.4) | 94.4 (39.8) | 119.4 (63.4)

OUTCOME MEASURES:

1. Primary Outcome: Count of Adverse Events Reported
Description: Measure reflects the total number of adverse events reported during course of the study.
Time Frame: Month 12
Measure: Number; unit: adverse events reported
Arm/Group | Arimoclomol | Placebo
Number analyzed (Participants) | 16 | 8
adverse events reported | 109 | 52

2. Secondary Outcome: Heat Shock Protein 70 (HSP70) Levels in the Tissue
Description: Biopsy taken from participants at baseline and month 4 visits. Measured change in HSP70 levels in the tissue.
Time Frame: Change from Baseline to Month 4
Measure: Mean (Standard Deviation); unit: ng/100ng myosin
Arm/Group | Arimoclomol | Placebo
Number analyzed (Participants) | 15 | 8
ng/100ng myosin | -110.72 (757.40) | -34.70 (336.35)

3. Secondary Outcome: Muscle Strength Testing
Description: Change in MMT score for the period. The MMT score range is 0-5. A score of 0 is the lowest and represents no visible or palpable contraction. A score of 5 is the highest and represents full range of motion against gravity, maximal resistance.
Time Frame: Change from Baseline to Month 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arimoclomol | Placebo
Number analyzed (Participants) | 15 | 8
units on a scale | -0.04 (0.19) | -0.12 (0.20)

4. Secondary Outcome: Muscle Strength Testing
Description: as for outcome 3
Time Frame: Change from Baseline to Month 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arimoclomol | Placebo
Number analyzed (Participants) | 13 | 8
units on a scale | -0.12 (0.22) | -0.26 (0.27)

5. Secondary Outcome: Muscle Strength Testing
Description: as for outcome 3
Time Frame: Change from Baseline to Month 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arimoclomol | Placebo
Number analyzed (Participants) | 14 | 7
units on a scale | -0.21 (0.21) | -0.35 (0.20)

6. Secondary Outcome: Inclusion Body Myositis-Functional Rating Scale (IBMFRS) Score
Description: Measured change for the period. The questionnaire has 10 questions. The maximum score is 40. The higher the score the better the functional status of the patient.
Time Frame: Change from Baseline to Month 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arimoclomol | Placebo
Number analyzed (Participants) | 16 | 8
units on a scale | -0.34 (1.38) | -0.88 (1.16)

7. Secondary Outcome: Inclusion Body Myositis-Functional Rating Scale (IBMFRS) Score
Description: as for outcome 6
Time Frame: Change from Baseline to Month 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arimoclomol | Placebo
Number analyzed (Participants) | 14 | 8
units on a scale | -0.68 (1.58) | -2.50 (3.31)

8. Secondary Outcome: Inclusion Body Myositis-Functional Rating Scale (IBMFRS) Score
Description: as for outcome 6
Time Frame: Change from Baseline to Month 12
Population: One of the subjects that dropped from the study in the Arimoclomol arm, returned for the 12 month visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arimoclomol | Placebo
Number analyzed (Participants) | 15 | 8
units on a scale | -2.03 (2.68) | -3.50 (3.35)

9. Secondary Outcome: Maximum Isometric Voluntary Contraction Testing (MVICT) Score
Description: Measured MVICT using the Quantitative Muscle Assessment (QMA) system designed by Computer Source, Atlanta, GA. The system uses an adjustable cuff to attach the patient's arm or leg to an inelastic strap that is connected to force transducer with a load of 0.5 to 1,000 Newtons. Maximum force is recorded.
Time Frame: Change from Baseline to Month 4
Measure: Mean (Standard Deviation); unit: newtons
Arm/Group | Arimoclomol | Placebo
Number analyzed (Participants) | 14 | 8
newtons | 0.46 (12.11) | -0.30 (14.49)

10. Secondary Outcome: Maximum Isometric Voluntary Contraction Testing (MVICT) Score
Description: as for outcome 9
Time Frame: Change from Baseline to Month 8
Measure: Mean (Standard Deviation); unit: newtons
Arm/Group | Arimoclomol | Placebo
Number analyzed (Participants) | 13 | 8
newtons | 7.20 (19.65) | -1.71 (17.80)

11. Secondary Outcome: Maximum Isometric Voluntary Contraction Testing (MVICT) Score
Description: as for outcome 9
Time Frame: Change from Baseline to Month 12
Measure: Mean (Standard Deviation); unit: newtons
Arm/Group | Arimoclomol | Placebo
Number analyzed (Participants) | 14 | 8
newtons | -1.21 (20.76) | 0.52 (17.98)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the subject's participation, 12 months.
Description: Participants were assessed at every study visit for adverse experiences. Safety laboratories were collected and monitored for all study participants.
Arm/Group | Arimoclomol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/8
Other Adverse Events (participants affected / at risk) | 16/16 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arimoclomol (N=16) | Placebo (N=8)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arimoclomol (N=16) | Placebo (N=8)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Dizziness/tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Dry eyes (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (4)
Throat irritation (Gastrointestinal disorders) | 3 (4) | 0 (0)
Loose stools (Gastrointestinal disorders) | 2 (2) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Painful parotids (Gastrointestinal disorders) | 0 (0) | 2 (2)
Bowel movement problems (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastralgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gas pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Geographic tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Loss of consciousness (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Sinus infection (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (4)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Leg ulcer infection (Infections and infestations) | 0 (0) | 1 (1)
Fall/contusion (Injury, poisoning and procedural complications) | 8 (23) | 5 (9)
Post-biopsy pain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Post-biopsy fatigue (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pruritus in biopsy scar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Finger cut (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyponatremia (Investigations) | 2 (2) | 0 (0)
High thyroxine levels (Investigations) | 1 (1) | 0 (0)
Spinal stenosis (Investigations) | 0 (0) | 1 (1)
Herniated disk (Investigations) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (10) | 2 (2)
Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis flare (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Heat and soreness of proximal lower limbs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (7) | 2 (3)
Worsening of restless leg syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Decreased libido (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Insect bite with erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cold sores (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 1 (1)
Sinus surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Solar lentigines removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 2 (3)
Edema (Vascular disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No